CLINICAL TRIAL: NCT06643858
Title: Establishment of Chinese Brain Charts for Individualized Diagnosis of Major Brain Diseases
Brief Title: Normal Chinese Lifespan Brain Charts Initiative (NCLBCI)
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Yaou Liu, Professor, Beijing Tiantan Hospital
Other Study IDs: KY2024-221-02
Record Dates: First submitted 2024-09-24; First posted 2024-10-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorders; Neurodegenerative Diseases; Cerebrovascular Diseases
Keywords: Brain Charts; Individualized Diagnosis
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Neurodegenerative Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nationwide retrospective neuroimaging data collection (5,000 participants): The primary imaging modalities include 3D T1-weighted imaging (3D T1WI) and 3D fluid-attenuated inversion recovery (3D FLAIR), along with basic demographic information, health status, and neuropsychological assessments.
  Interventions: Other: No intervention
- Nationwide prospective neuroimaging cohort of the Chinese normal population (5,000 participants).: This cohort will include multimodal imaging sequences (3D T1-weighted imaging, 3D FLAIR, diffusion kurtosis imaging [DKI], arterial spin labeling [ASL], vascular water exchange imaging [VEXI], magnetic resonance angiography [MRA], and resting-state functional MRI [rest-fMRI]). Detailed demographic information, neuropsychological assessments, standardized questionnaires, and basic physical examinations will also be collected. Multimodal neuroimaging data and neuropsychological assessments will be followed up twice (at 1 year and 2 years).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study does not involve any interventions.

SUMMARY:
Major brain diseases (including neuroimmune diseases, neurodegenerative diseases, and cerebrovascular diseases) are leading causes of death and disability in humans. This research will gather brain imaging data from more than 10,000 participants across multiple age groups from multiple centers nationwide. Using standardized modeling methods, the investigators aim to establish normal brain imaging reference values for the Chinese population. (1) The study will reveal population-level patterns of brain structure changes and determine normal reference values for brain structure at different ages. (2) Non-invasive imaging methods will be applied to evaluate blood-brain barrier changes without the need for invasive procedures, establishing age-related permeability patterns and normal values in healthy populations. Additionally, functional magnetic resonance imaging (fMRI) will be combined to provide brain function indicators at various scales, creating comprehensive multi-dimensional function charts. (3) These brain structure and function charts will be applied to the individualized diagnosis and treatment of major brain diseases, including neuroimmune diseases (Multiple Sclerosis [MS], Neuromyelitis Optica Spectrum Disorders [NMOSD]), neurodegenerative diseases (Alzheimer's disease [AD], Parkinson's disease [PD]), and cerebrovascular diseases (Cerebral Small Vessel Diseases [cSVD]). This approach will facilitate early disease diagnosis and provide precise, individualized assessments of treatment efficacy and prognosis prediction. The established brain structure and function charts will be accessible via interactive websites or software, enabling real-time online data updates and individualized percentile outputs for brain structure and function. By inputting the target data, users can obtain individualized evaluation metrics for brain structure and function. The project's implementation and application hold great potential for broad use, promotion, and high translational potential.

DETAILED DESCRIPTION:
In 2022, the World Health Organization (WHO) issued a policy document calling for attention to brain health and neurological diseases. In China's "14th Five-Year Plan," brain science research is designated as one of the key research areas, with the development goal of promoting the understanding of fundamental brain mechanisms and meeting the needs for improving brain health in the population. Understanding brain development and aging in healthy individuals is a prerequisite for comprehending neurological diseases. The function of the blood-brain barrier is crucial to maintaining brain health and plays a central role in the occurrence and development of major brain diseases. However, there is currently a lack of standardized reference values for brain structural imaging evaluation, and even less is known about the changes in blood-brain barrier function in healthy populations. This significantly hinders the understanding of brain health, the pathology of major brain diseases, and the ability to make early individualized diagnoses and treatments. Additionally, although functional Magnetic Resonance Imaging (fMRI) has become an essential research tool in neuroscience, its clinical application is still fraught with difficulties, primarily due to the lack of standardized quantitative evaluation methods. In 2022, international datasets covering the human lifespan were established, and the constructed percentile curves revealed population patterns of brain development and individualized differences, offering a promising standardized tool for evaluating brain health and diseases. Nevertheless, existing brain imaging characterizations still have some limitations: (1) the lack of normal reference values for brain imaging structures in the Chinese population; (2) the absence of brain function indicator charts, such as functional connectivity and cerebral blood flow perfusion, especially with regard to the critical role of blood-brain barrier changes in major brain disease transformation; (3) The application value of brain charts in the diagnosis and treatment of major brain diseases lacks systematic research. Therefore, constructing brain structure and function imaging charts (normal reference values) for the Chinese population is imperative and represents a pressing scientific and clinical issue that needs to be addressed.

Establishment of the Chinese Normal Population Neuroimaging Database: The investigators aim to establish the largest neuroimaging research cohort in China, consisting of 10,000 participants, with a wide age range (6-90 years), balanced gender distribution, and representation from more than 30 centers nationwide, ensuring a balanced distribution of scanning devices. Using federated machine learning methods, the study will address data privacy and security concerns. This project primarily includes: ① Retrospective collection of neuroimaging data from 5,000 participants nationwide, focusing mainly on 3DT1WI and 3DFLAIR imaging, and also collecting basic demographic information, health status, and neuropsychological assessments. ② A prospective neuroimaging cohort of 5,000 participants from the Chinese normal population, including multimodal imaging sequences (3DT1WI, 3DFLAIR, DKI, ASL, VEXI, MRA, and resting-state fMRI), along with detailed demographic information, neuropsychological assessments, standardized questionnaires, and basic physical examinations. Multimodal neuroimaging data and neuropsychological assessments will be collected at two follow-ups (1-year and 2-year intervals). Among the multimodal brain imaging collected, the method reflecting blood-brain barrier permeability is vascular water exchange MRI (VEXI), which uses water molecules as natural internal tracers to measure blood-brain barrier function.

Establishment of Brain Structure and Function Charts for the Chinese Normal Population: Based on retrospective and prospective neuroimaging data from the Chinese normal population, standardized modeling methods (including Generalized Additive Mixed Models [GAMLSS] and Gaussian Process Regression [GPR]) will be used to create structural brain charts. These charts will include: ① Whole brain volumes (Gray Matter Volume [GMV], White Matter Volume [WMV], Total Intracranial Volume [TIV], etc.), the volumes of 148 brain regions, and subcortical nuclei volumes. ② White matter fiber tracts (48 white matter fiber tracts and diffusion metrics, including Fractional Anisotropy [FA], Mean Kurtosis [MK], Mean Diffusivity [MD], etc.) and functional brain charts, which include: ① Blood-brain barrier permeability; ② Cerebral blood flow (CBF); ③ Local brain activity indicators (Regional Homogeneity [ReHo], Amplitude of Low-Frequency Fluctuations [ALFF], etc.); ④ Global functional connectivity; and ⑤ Brain network analysis (local and global efficiency), among others.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals with normal physical function who can lie supine without medical issues (e.g., no difficulty breathing, physical pain, nausea, or dizziness);
2. No claustrophobia;
3. No metal implants in the body (e.g., metal teeth, intrauterine devices, pacemakers, etc.).

Exclusion Criteria:

1. Presence of metal implants in the body;
2. Individuals who have undergone aneurysm surgery or have aneurysm clips in the brain;
3. Contraindications to MRI examination;
4. Prospective cohort participants who are unable to meet follow-up requirements.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy individuals aged 6 to 90 years are eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Brain Imaging Scans Collected and Processed Across Multiple Centers | December 2023 - May 2025
  The primary outcome will be the total number of brain imaging scans (including 3DT1WI, 3DFLAIR, DKI, ASL, VEXI, MRA, and resting-state fMRI) successfully collected and processed across multiple centers. These scans will be aggregated by type (e.g., 3DT1WI, 3DFLAIR) and by imaging modality. Standardized imaging processing methods will be applied to ensure consistency in data quality and preparation for constructing brain structure and function charts.
Accuracy and Reliability of Structural Brain Chart Models | December 2023 - November 2025
  The primary outcome will be the accuracy and reliability of the structural brain chart models, assessed through metrics such as mean absolute error (MAE), R-squared (R²), and Z-scores across multiple centers. Model performance will be evaluated based on the deviation of predicted brain structure volumes (e.g., gray matter volume, white matter volume, total intracranial volume) from actual collected data. Validation will include testing the charts on retrospective and prospective datasets from the primary center and additional participating centers. The models will be optimized iteratively based on these evaluations.
Accuracy and Reliability of Functional Brain Chart Models | December 2024 - May 2026
  The outcome will be the accuracy and reliability of the functional brain chart models, assessed using metrics such as correlation coefficients, Z-scores, and functional connectivity strength across multiple brain regions. The performance will be validated using longitudinal multimodal functional brain data (e.g., resting-state fMRI, cerebral blood flow, regional homogeneity). Model reliability will be evaluated by comparing predicted functional measures with observed data across longitudinal time points.
User Access and Interaction Metrics on Brain Chart Online Platform | June 2025 - May 2026
  The outcome will measure the number of user interactions and successful use cases on the real-time interactive online platform. Key metrics will include the number of users, frequency of data input and retrieval, and the accuracy of the generated individualized brain structure and function parameters based on user-provided data. Platform reliability and performance will be validated through user feedback and system testing.
Number of Brain Chart Products Released and Marketed | June 2026 - November 2026
  The outcome will measure the number of brain chart products that have been successfully productized and promoted for market application. This includes the completion of product development, official product launches, and market penetration metrics such as user adoption rates and commercial distribution.

SECONDARY OUTCOMES:
Number of Peer-Reviewed Papers Published and Patents Filed | June 2024 - November 2026
  The outcome will be the total number of peer-reviewed scientific papers published (targeting 3-4) and the number of national invention patents filed (targeting 5-7). This includes metrics for the quality of journals (impact factors) and patent filing stages (application, approval).
Number of Multicenter Sites Using Brain Charts for Clinical and Research Purposes | December 2025 - November 2026
  The outcome will measure the number of additional multicenter sites that have adopted and integrated the brain charts into their clinical and research workflows. This will include the number of sites actively participating in ongoing validation and refinement of the brain charts, with metrics for data sharing, collaboration, and feedback implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Yaou Liu, Doctor, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Clinical and MR data can be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 3 years after the end of the trial.
Access Criteria: The neurosurgeon and radiologist submitting the application to Professor Liu.